CLINICAL TRIAL: NCT05596396
Title: Feasibility and Acceptability of a Guided E-health Program (LifeHack), With and Without a Fixed Structure, to Improve Well-being in University Students.
Brief Title: The Caring Universities Project: LifeHack
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: VU University of Amsterdam (Other)
Collaborators: Erasmus University Rotterdam (Other); University of Amsterdam (Other); Leiden University (Other); Maastricht University (Other); Utrecht University (Other); InHolland University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Arpana Amarnath, Research Associate, VU University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VCWE-2021-175
Record Dates: First submitted 2022-10-12; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Well-being
Keywords: well-being; positive mental health; guided; e-health; university students

STUDY DESIGN:
Intervention Model Description: The present study is a two-armed randomized controlled trial. This trial will be conducted in a university setting. A guided web-based intervention to improve positive mental health and well-being (LifeHack) will be compared to an unstructured version of the same intervention (LifeHack-C)
Who Masked: Investigator, Outcomes Assessor
Masking Description: An independent researcher who is not involved in the study will generate the random sequence using a computer random sequence generator. Randomisation will take place at an individual level, stratified by gender and the university where students study. Participants will be randomised into two groups (LifeHack vs LifeHack-C) with an allocation ratio of 1:1. Block randomisation with randomly varied block sizes (6 to 12 allocations per block) will be conducted to prevent foreknowledge of intervention assignment. Allocation will be concealed from the study's researchers. It is not possible to mask personnel and participants to the treatment allocation because of the nature of the intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LifeHack (Experimental): Participants assigned to this arm will receive a 6-week guided e-health intervention to increase positive mental health and well-being.
  Interventions: Behavioral: LifeHack
- LifeHack-C (Active Comparator): Participants assigned to this arm will receive the same intervention, delivered over 2 to 6 weeks.
  Interventions: Behavioral: LifeHack-C

INTERVENTIONS:
Behavioral: LifeHack — Participants assigned to LifeHack will follow a six week-guided online intervention with a fixed structure where the themes are delivered in a predefined order, and the contents get unlocked sequentially. The first mandatory module is the introduction module which also functions as a goal-setting module. Following this, students complete one mandatory module per week (and the optional modules if they choose to do so) delivered sequentially, starting with the theme of mood, studies, social life and finally, self-esteem. Students complete the themes one by one and the consecutive themes (and modules) are unlocked only after completing the main module of the assigned theme.
  Arms: LifeHack
Behavioral: LifeHack-C — Participants assigned to LifeHack-C will receive the same guided online intervention, but they can choose what theme they would like to start with, when to work on it and how many modules they wish to complete. After completing the introduction module, the participants will be advised to complete two modules per week and at least four in total. Therefore, the program's duration will be approximately two and six weeks. However, participants can follow the program at their own pace.
  Arms: LifeHack-C

SUMMARY:
Within the Caring Universities project (study protocol VCWE- 2021-175 accepted by the VCWE), the investigators have developed a guided e-health programme (LifeHack) designed to improve positive mental health in university students. With the current study, the investigators aim to examine the feasibility and acceptability of LifeHack - with and without a fixed structure - to improve students' positive mental health and well-being.

The secondary goals are to gain insight into pre-test to post-test differences regarding general well-being, symptoms of depression, anxiety and quality of life.

DETAILED DESCRIPTION:
The present study is a two-armed randomized controlled trial. This trial will be conducted in a university setting. Participants will be randomized to receive a version of the intervention either with a fixed structure (LifeHack) or a flexible structure (LifeHack-C).

LifeHack was developed based on existing literature and adapted in collaboration with university students to meet the specific needs of the university students. LifeHack is based on cognitive-behavioural therapy (CBT). It consists of fourteen modules, of which six are principal (compulsory) modules. These include one introductory module, four main modules covering the themes of mood, studies, social life and self-esteem, and one closing module. In addition, there are two optional modules per theme, totalling to eight optional modules.

Every module consists of evidence-based information, exercises, and homework assignments that are delivered via computer, laptop, tablet, or mobile phone. The content is delivered in text format with pictures and infographics. The intervention is available in both English and Dutch.

Participants assigned to LifeHack will follow a fixed structure where the themes are delivered in a predefined order, and the contents get unlocked sequentially. Participants assigned to LifeHack-C will receive the same intervention, but they can choose what theme they would like to start with, when to work on it and how many modules they wish to complete.

Every week trained e-coaches (trained clinical psychology master students) will provide asynchronous written personalized feedback to each participant on the progress of the program and the exercises via the program platform. Measurements include post-test assessment of adherence, treatment satisfaction, and satisfaction with e-coach. Secondary outcomes include pre and post-assessment of well-being, common measures of psychopathology symptoms, and quality of life.

Data will be analysed based on the intent to treat principle.

All students currently enrolled at the participating universities (Vrije Universiteit Amsterdam, Erasmus University, InHolland University of Applied sciences, Universities of Amsterdam, Leiden, Utrecht and Maastricht) are potentially eligible for the trial.

Students can participate in LifeHack free of charge, which will likely improve their general well-being. They will not receive any additional incentives for participation.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this trial, a subject must meet all the following criteria:

* Being fluent in Dutch and/or English
* Being enrolled as a student of the seven participating universities
* Being 16 years of age or older
* Having access to a PC or mobile device with internet access
* Provide informed consent before participation

Exclusion Criteria:

* None. All interested students are eligible to participate.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with the intervention | T1 (post test: 4-weeks)
  The Client Satisfaction Questionnaire (CSQ-8) is used to measure participants' satisfaction with the overall intervention. The CSQ-8 is commonly used to measure satisfaction with online interventions. It consists of eight items on a four-point Likert scale with a total score ranging from 8 to 32, where a higher score indicates greater satisfaction.
Treatment Adherence | T1 (post test: 4-weeks)
  Adherence refers to the degree to which the user followed the program as it was designed. The present study measures adherence by dividing the number of modules completed by a participant at the time of post-test by the total number of modules in the programme and multiplying this by 100. The resulting percentage will indicate the completion rate.
Satisfaction with E-coach | T1 (post test: 4-weeks)
  The Working Alliance Inventory for guided internet interventions (WAI-I) is used to evaluate participant's satisfaction with the e-coach. The WAI-I consists of 12 items on a 5-point Likert scale with a total score ranging from 12 to 60, where higher scores indicate higher satisfaction
Usability | T1 (post test: 4-weeks)
  The System Usability Scale (SUS-10) is used to measure the usability of the intervention. It consists of 10 items on a five-point Likert scale with a total score ranging from 0 to 100, where a higher score indicates greater usability.

SECONDARY OUTCOMES:
Change in positive mental health and well-being | T0 (Baseline) to T1 (Post-test: 4-weeks)
  The Mental Health Continuum - Short Form (MHC-SF) is used to measure positive mental health. It comprises of 14 items that represent various feelings of emotional, psychological and social well-being. These items are measured on a six point Likert scale ranging from 1 (never) to 6 (every day). The scores range from 14 to 84 with higher scores indication greater positive mental health and well-being.
Change in depressive symptoms | T0 (Baseline) to T1 (Post-test: 4-weeks)
  The Patient Health Questionnaire (PHQ-9) is used as the measure of depression. This questionnaire consists of 9 items scored on a four-point Likert scale ranging from 0 (not at all) to 3 (nearly every day). The total scores can range from 0 to 27, with higher scores indication more severe depressive symptoms.
Change in Anxiety symptoms | T0 (Baseline) to T1 (Post-test: 4-weeks)
  The Generalized Anxiety Disorder scale (GAD-7) is used to measure symptoms of generalized anxiety. The questionnaire consists of 7 items measured on a four-point Likert ranging from 0 (not at all) to 3 (nearly every day). The total scores range from 0 to 21 with higher scores indicating more severe GAD symptoms.

OTHER OUTCOMES:
Socio demographic characteristics of participants | T0 (Baseline)
  age, gender, ethnicity, student status, study level, relationship status, whether the student is currently undergoing any treatment (pharmacotherapy/psychotherapy/both/none)
Satisfaction with individual modules | After completing each module, through Week 1, Week 2, Week 3, Week 4
  After completing each module, the participants respond to the question "how useful was this module" on a scale of 1 - 100, with higher scores indicating better satisfaction with the module.

CONTACTS AND LOCATIONS:
Overall Officials: Pim Cuijpers, dr. Prof, Study Director — VU University of Amsterdam
Locations (1):
- Vrije Universiteit Amsterdam, Amsterdam, Netherlands